CLINICAL TRIAL: NCT02687828
Title: A Prospective, Mono-Country and Multi-center Study to Observe Safety and Effectiveness of Adalimumab in KoREan Intestinal Behcet's Disease(BD) Patients
Acronym: AMORE
Status: Completed | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P15-760
Record Dates: First submitted 2016-02-17; First posted 2016-02-22 (Estimated); Last update posted 2021-03-22 (Actual); Status verified 2021-03

CONDITIONS: Intestinal Behcet's Disease (BD)
Keywords: Intestinal Behcet's disease (BD); Adalimumab; Safety; Effectiveness; AMORE study

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Subjects receiving adalimumab: The subjects who are prescribed adalimumab for intestinal Behcet's disease (BD) in accordance with the approved Korean label.

SUMMARY:
This study evaluates the safety profile and effectiveness of adalimumab in Korean intestinal Behcet's disease (BD) patients in routine clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be an adult >= 19 years
* Subjects who are eligible to be treated with adalimumab for intestinal Behcet's disease in accordance with the approved label in Korea
* Subjects provide written authorization form for use/disclose of personal health data prior to participating in this study

Exclusion Criteria:

* Subjects who are contraindicated to any anti-TNF agent
* Female subjects who are pregnant or breast feeding
* Subjects who are participating in other interventional clinical trials

Ages: 19 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Intestinal Behcet's disease (BD) patients who are eligible to be prescribed adalimumab by the treating investigator as per Korean label will be enrolled.
Sampling Method: Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2016-02-18 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events | From Day 1 to 70 days following 56 weeks from first dose of adalimumab or the last administration of adalimumab if the participant stopped receiving adalimumab before 56 weeks
  All adverse events including serious and unexpected events will be assessed.

SECONDARY OUTCOMES:
Number of participants with adverse drug reactions | From Day 1 to 70 days following 56 weeks from first dose of adalimumab or the last administration of adalimumab if the participant stopped receiving adalimumab before 56 weeks
  All adverse reactions including serious and unexpected reactions will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie
Locations (10):
- South Korea (10):
  - Kyungpook National Univ Hosp /ID# 147937, Daegu, Daegu Gwang Yeogsi
  - Ajou University Hospital /ID# 147938, Suwon, Gyeonggido
  - Pusan Nat Univ Yangsan Hosp /ID# 169243, Yangsan, Gyeongsangnam-do
  - Yonsei University Health System, Severance Hospital /ID# 147932, Seodaemun-gu, Seoul Teugbyeolsi
  - Samsung Medical Center /ID# 147934, Seoul, Seoul Teugbyeolsi
  - Cath Univ Seoul St Mary's Hosp /ID# 147936, Seoul, Seoul Teugbyeolsi
  - Kosin University Gospel Hosp /ID# 169244, Busan
  - The Catholic Univ. of Korea /ID# 169245, Gyeonggi-do
  - Seoul National University Hospital /ID# 147933, Seoul
  - Asan Medical Center /ID# 147935, Seoul

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: clinical study report synopsis — https://www.abbvie.com/content/dam/abbvie-dotcom/clinical-trials/adalimumab_P15-760.pdf